CLINICAL TRIAL: NCT00596427
Title: Effects of Colesevelam HCl on Hepatic Insulin Sensitivity, Gluconeogenesis, Glucose Absorption and Lipid Synthesis in Subjects With Type 2 Diabetes Mellitus
Brief Title: Mechanisms of Glucose Lowering Effect of Colesevelam HCl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carine Beysen (Industry)
Responsible Party: Sponsor-Investigator, Carine Beysen, Director, Clinical Metabolic Research, KineMed
Organization: KineMed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KM-11A
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes
Keywords: type two diabetes; gluconeogenesis; glucose; lipid synthesis; hepatic insulin sensitivity; colesevelam HCl
MeSH Terms: conditions — Diabetes Mellitus | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo tablet 3 tablets 2x/day (Placebo Comparator): Type-2 diabetes mellitus patients
  Interventions: Drug: Placebo
- Colesevelam HCL 625 mg: 3 tablets 2x/day (Experimental): Type-2 diabetes mellitus patients
  Interventions: Drug: Colesevelam HCL

INTERVENTIONS:
Drug: Colesevelam HCL — Colesevelam HCL 625 mg: 3 tablets twice per day
  Other Names: WelChol
  Arms: Colesevelam HCL 625 mg: 3 tablets 2x/day
Drug: Placebo — Placebo tablets: 3 tablets twice per day
  Arms: Placebo tablet 3 tablets 2x/day

SUMMARY:
The mechanism by which colesevelam HCl lowers glucose is not known. Knowledge of the potential mechanism of action is important for defining the role of the drug among oral antidiabetic agents available for use in subjects with diabetes. The objective of this study is to provide insight into the mechanisms of action of colesevelam HCl in T2DM. The mechanisms of interest include hepatic insulin sensitivity, rate of appearance of exogenous glucose and changes in incretin hormone concentrations.

DETAILED DESCRIPTION:
Colesevelam HCl (marketed in the U.S. as WelChol®) is a non-absorbed polymer that binds bile acids in the intestine, impeding their reabsorption, and is indicated to lower low-density lipoprotein cholesterol (LDL-C) in subjects with hypercholesterolemia. As the bile acid pool becomes depleted, the hepatic enzyme cholesterol 7-(alpha)-hydroxylase is upregulated, increasing the conversion of cholesterol to bile acids. This causes an increased demand for cholesterol in the liver, resulting in the dual effect of increasing transcription and activity of the cholesterol biosynthetic enzyme, hydroxymethyl-glutaryl-coenzyme A (HMG CoA) reductase, and increasing the number of hepatic low-density lipoprotein (LDL) receptors. These compensatory effects increase the clearance of LDL-C from the blood, decreasing serum LDL C levels (1; 2).

Recently, it has been shown that colesevelam HCl also improves glycemic control in subjects with T2DM who are not controlled adequately on metformin, sulfonylurea or a combination of the two drugs (3). The mechanism of action for glucose lowering is not known. Improved glycemic control with colesevelam HCl treatment could be due to any of several mechanisms. Colesevelam HCl could reduce hepatic insulin resistance and lead to a decrease in hepatic glucose production (HGP). The observation by Schwartz et al (4) of significantly reduced fasting plasma glucose concentrations in colesevelam-treated T2DM patients suggests such a reduction in HGP, as fasting hyperglycemia is a direct function of HGP. Colesevelam HCl could also decrease post-prandial glucose absorption. Changes in glucose absorption with other bile acid sequestrants (BAS) (5) and bile acids (6) have been reported.

With regard to molecular mediators of the colesevelam effect on glucose metabolism, there is considerable evidence emerging about the role of bile acids and nuclear transcription factors, such as the farnesyl X receptor (FXR), in the regulation of glucose and lipid metabolism (7) (8) (9-15). Changes in cellular lipids or nuclear hormone receptors might directly alter HGP although mechanisms leading to changes in hepatic lipid and glucose metabolism by colesevelam HCl have not previously been investigated.

Significant changes in cholesterol and bile acid synthesis rates are expected with colesevelam treatment. BAS treatment can alter the transhepatic flux and compositional profile of the circulating bile acid pool (16), and thus its hydrophobicity, and this may effect the activation of nuclear receptors, including FXR (17; 18). Determination of the effect of colesevelam treatment on bile acid synthesis may provide evidence for its metabolic effects. The effects on hepatic fatty acid synthesis (de novo lipogenesis or DNL) have not been investigated and may provide further evidence for a metabolic effect of colesevelam.

Specific hypotheses about its mode of action will be tested, focusing on hepatic glucose metabolism and intestinal glucose absorption.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria at the Screening Visit will be eligible to participate in the trial:

* Have given written informed consent
* Male or Female

  1. Females of childbearing potential who are on approved birth control method:

     oral, injectable, or implantable hormonal contraceptives; intrauterine device; diaphragm plus spermicide or female condom plus spermicide
  2. Females of non-childbearing potential: hysterectomy, tubal ligation 6 months prior screening or post-menopausal for at least 1 year
* Previously diagnosed or newly diagnosed with T2DM
* Age 30 to 70 years, inclusive
* BMI ≥ 18.5 kg/m2 and ≤ 40 kg/m2
* HbA1C 7-10%, inclusive (exceptions between 6.7-7% may be enrolled with prior approval of SPONSOR)
* Fasting plasma glucose < 300 mg/dL
* Diet controlled or on stable dose of a sulfonylurea and/or meglitinides and/or metformin for ≥ 90 days before screening
* No history of liver, biliary or intestinal disease (AST/ALT < 2X upper limit of normal value)
* Normal TSH
* Agrees to maintain their regular diet and exercise routine
* Agrees to refrain from consumption of alcohol 48 hours prior to start of infusions (week 0 and week 12)

Exclusion Criteria:

Subjects are excluded from participation in the study if any of the following criteria apply:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Treatment with lipid lowering medication other than statins
* Treatment with statins that have not been stable for 3 months before screening
* Treatment with colesevelam HCl, cholestyramine or colestipol for hyperlipidemia within the last 3 months of screening
* Treatment with a thiazolidinedione (TZD) at any time
* Treatment with acarbose at any time
* Treatment with insulin in the past 6 months
* Treatment with antibiotics within the last 3 months
* Treatment with any medication affecting liver or intestinal function within the last 3 months
* Pregnant
* Breastfeeding
* Has had unstable weight within the last 3 months of screening (± 5 kg)
* History of an allergic or toxic reaction to colesevelam HCl
* History of dysphagia, swallowing disorders, or intestinal motility disorder
* Serum triglycerides ≥ 350 mg/dL at screening visit (exceptions up to 500 mg/dl may be enrolled with prior approval of SPONSOR)
* Serum LDL-C <60 mg/dL at screening visit
* Any condition or therapy which, in the opinion of the investigator, poses a risk to the subject or makes participation not in the subject's best interest
* Use of any investigational drug within 3 months of screening
* Chronic treatment with oral corticosteroids at any time or acute treatment within the last 3 months
* History of drug or alcohol abuse, is currently a user (including "recreational use") of any illicit drugs, or has a positive urine drug screen at screening
* Donated a unit of blood within 30 days before screening

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Beysen, PhD, Principal Investigator — KineMed
Locations (3):
- United States (3):
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Clinical Pharmacology of Miami, Inc, Miami, Florida
  - Diabetes & Glandular Disease Research Associates, San Antonio, Texas

REFERENCES:
- [Background] Grundy SM, Ahrens EH Jr, Salen G. Interruption of the enterohepatic circulation of bile acids in man: comparative effects of cholestyramine and ileal exclusion on cholesterol metabolism. J Lab Clin Med. 1971 Jul;78(1):94-121. No abstract available. PMID 5569253
- [Background] Shepherd J, Packard CJ, Bicker S, Lawrie TD, Morgan HG. Cholestyramine promotes receptor-mediated low-density-lipoprotein catabolism. N Engl J Med. 1980 May 29;302(22):1219-22. doi: 10.1056/NEJM198005293022202. PMID 7366673
- [Background] Zieve FJ, Kalin MF, Schwartz SL, Jones MR, Bailey WL. Results of the glucose-lowering effect of WelChol study (GLOWS): a randomized, double-blind, placebo-controlled pilot study evaluating the effect of colesevelam hydrochloride on glycemic control in subjects with type 2 diabetes. Clin Ther. 2007 Jan;29(1):74-83. doi: 10.1016/j.clinthera.2007.01.003. PMID 17379048
- [Background] Jenkins DJ, Wolever TM, Leeds AR, Gassull MA, Haisman P, Dilawari J, Goff DV, Metz GL, Alberti KG. Dietary fibres, fibre analogues, and glucose tolerance: importance of viscosity. Br Med J. 1978 May 27;1(6124):1392-4. doi: 10.1136/bmj.1.6124.1392. PMID 647304
- [Derived] Beysen C, Murphy EJ, Deines K, Chan M, Tsang E, Glass A, Turner SM, Protasio J, Riiff T, Hellerstein MK. Effect of bile acid sequestrants on glucose metabolism, hepatic de novo lipogenesis, and cholesterol and bile acid kinetics in type 2 diabetes: a randomised controlled study. Diabetologia. 2012 Feb;55(2):432-42. doi: 10.1007/s00125-011-2382-3. Epub 2011 Dec 2. PMID 22134839
- See also: KineMed, Inc. — http://www.kinemed.com
- See also: Diablo Clinical Research, Inc. — http://www.diabloclinical.com/
- See also: WelChol — http://www.welchol.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with type 2 diabetes. All pre-existing drug treatments were stable for at least 3 months prior.
Pre-assignment Details: Participants excluded based on fasting plasma glucose levels, fasting serum triglyceride levels, LDL-cholesterol levels, pregnancy or a history of liver, biliary, or intestinal diseases. Participants treated with insulin or lipid agent less than six months prior were excluded as well.
Groups:
- Type-2 Diabetes Mellitus Patients Treated With Colesevelam: Subjects received six tablets a day of colesevelam (3.75g/day) for 12 weeks; three tablets with lunch and three tablets with dinner.
- Type-2 Diabetes Mellitus Patients Treated With Placebo: Subjects received six tablets a day of matched placebo(3.75g/day) for 12 weeks; three tablets with lunch and three tablets with dinner.
Period: Overall Study
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Started | 30 | 30
Completed | 26 | 28
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Increased Fasting Triacylglycerol level | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 6 | 5 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (9) | 56 (9) | 57.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 18 | 16 | 34
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
BMI [Mean (Standard Deviation); unit: kg/m2] — Baseline participant characteristics.
  kg/m2 | 30 (5) | 31 (5) | 30.5 (5)
Weight [Mean (Standard Deviation); unit: kg] — Baseline participant characteristics.
  kg | 84 (16) | 88 (19) | 86 (18)
HbA 1c [Mean (Standard Deviation); unit: percentage] | 8.5 (1.2) | 8.0 (0.9) | 8.25 (1.05)
Glucose [Mean (Standard Deviation); unit: mmol/l] | 9.2 (2.3) | 8.4 (2.4) | 8.8 (2.3)
Insulin [Mean (Standard Deviation); unit: pmol/l] | 76 (42) | 97 (42) | 87 (42)
Total cholesterol [Mean (Standard Deviation); unit: mmol/l] | 4.6 (1.2) | 4.6 (1.3) | 4.6 (1.3)
LDL-cholesterol [Mean (Standard Deviation); unit: mmol/l] | 2.8 (0.8) | 2.8 (1.0) | 2.8 (0.9)
HDL-cholesterol [Mean (Standard Deviation); unit: mmol/l] | 0.9 (0.2) | 1.0 (0.2) | 1.0 (0.2)
Triacylglycerol [Mean (Standard Deviation); unit: mmol/l] | 2.2 (0.8) | 2.0 (0.9) | 2.1 (0.9)

OUTCOME MEASURES:

1. Secondary Outcome: Total Glucagon-like Peptide (GLP-1) Area Under the Curve (AUC)
Description: Changes from baseline of total GLP-1 AUC after 12 weeks of placebo or colesevelam treatment.
  AUC values were calculated by the trapezoid method using all results between 0 and 300 minutes
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: picomoles (pmol)/Liter (L) x minute (min
Groups:
- Type-2 Diabetes Mellitus Patients Treated With Placebo: Subjects received six tablets a day of colesevelam matched placebo for 12 weeks; three tablets with lunch and three tablets with dinner.
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
picomoles (pmol)/Liter (L) x minute (min | 5 (2) | -3 (1)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Change from baseline between groups were compared; Test type: Superiority or Other; p < 0.01, mixed-effects regression models

2. Secondary Outcome: Total Glucose-dependent Insulinotropic Polypeptide (GIP) AUC
Description: Changes from baseline of total GIP-1 AUC after 12 weeks of placebo or colesevelam treatment.
  AUC values were calculated by the trapezoid method using all results between 0 and 300 minutes
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/l x min
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
pmol/l x min | 7 (2) | -6 (2)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Change from baseline between groups was compared; Test type: Superiority or Other; p < 0.001, mixed-effects regression models

3. Primary Outcome: Fasting Endogenous Glucose Production (EGP)
Description: Changes from baseline of fasting EGP after 12 weeks of placebo or colesevelam treatment.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: umol per kg Fat-Free Mass (FFM) per min
Groups:
- Type-2 Diabetes Mellitus Patients Treated With Colesevelam: Subjects received six tablets a day of colesevelam (3.75grams/day) for 12 weeks; three tablets with lunch and three tablets with dinner.
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 27
umol per kg Fat-Free Mass (FFM) per min | 0.19 (0.78) | 1.59 (0.77)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Comparison of change from baseline between groups (treatment effect); Test type: Superiority or Other; p < 0.1, mixed-effects regression models; This model had fixed effects of treatment, visit and treatment by visit interaction and a random subject effect

4. Other Pre Specified Outcome: Glycosylated Hemoglobin (HbAlc)
Description: Changes from baseline of HbA1c after 12 weeks of placebo or colesevelam treatment.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
percentage | -0.3 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Test type: Superiority or Other; p < 0.01, mixed-effects regression models

5. Other Pre Specified Outcome: Glucose AUC
Description: Changes from baseline of glucose AUC after 12 weeks of placebo or colesevelam treatment.
  AUC values were calculated by the trapezoid method using all results between 0 and 300 minutes
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: millimoles (mmol)/l x min
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
millimoles (mmol)/l x min | -0.8 (0.4) | 0.5 (0.4)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Test type: Superiority or Other; p < 0.05, mixed-effects regression models

6. Primary Outcome: Fasting Gluconeogenesis
Description: Change from baseline of fasting gluconeogenesis after 12 weeks of placebo or colesevelam treatment.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: micromoles (µmol) per kg FFM per min
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 26
micromoles (µmol) per kg FFM per min | 0.02 (0.32) | -0.19 (0.27)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Change from baseline between groups were compared (treatment effect); Test type: Superiority or Other; p < 0.1, mixed-effects regression models

7. Primary Outcome: Fasting Glycogenolysis
Description: Change from baseline of fasting glycogenolysis after 12 weeks of placebo or colesevelam treatment.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: µmol per kilograms (kg) FFM per min
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 25
µmol per kilograms (kg) FFM per min | 0.11 (0.81) | 1.78 (0.69)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Test type: Superiority or Other; p = 0.05, mixed-effects regression models

8. Primary Outcome: Rate of Appearance of Exogenous Glucose (Glucose Absorption)
Description: Change from baseline of the rate of appearance of oral glucose after 12 weeks of placebo or colesevelam treatment. Mean of values obtained between 0 and 300 min is reported.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: µmol per kg FFM per minute (min)
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 25 | 26
µmol per kg FFM per minute (min) | 0 (0.56) | 1 (0.63)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Test type: Superiority or Other; p = 0.6, mixed-effects regression models

9. Secondary Outcome: Fasting Fractional De Novo Lipogenesis (DNL)
Description: Changes from baseline in fasting fractional DNL after 12 weeks of colesevelam or placebo treatment were calculated. Fractional DNL represents the fraction of palmitate in very-low density lipoproteins-triglycerides (VLDL-TG) that was newly synthesized.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: percent new palmitate
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 26
percent new palmitate | -0.6 (0.57) | -1.4 (0.58)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam; Treatment effect of change from baseline; Test type: Superiority or Other; p = 0.3, mixed-effects regression models

10. Secondary Outcome: Fasting Fractional Cholesterol Synthesis
Description: Changes from baseline in fasting fractional cholesterol synthesis after 12 weeks of colesevelam or placebo treatment. Fractional Cholesterol synthesis represents the fraction of free cholesterol in plasma that was newly synthesised.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: Percent new cholesterol
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
Percent new cholesterol | 3.0 (0.4) | 0.5 (0.4)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam; Treatment effect of change from baseline; Test type: Superiority or Other; p < 0.0001, mixed-effects regression models

11. Secondary Outcome: Postprandial Fractional Cholic Acid Synthesis
Description: Changes from baseline in fractional cholic acid synthesis after 12 weeks of colesevelam or placebo treatment were evaluated. Fractional cholic acid synthesis represents the relative amount of cholic acid that is made from newly synthesised cholesterol.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: Percent new cholic acid
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
Percent new cholic acid | 5.5 (1.0) | 1.7 (1.0)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam; Treatment effect of change from baseline; Test type: Superiority or Other; p < 0.01, mixed-effects regression models

12. Secondary Outcome: Glucagon AUC
Description: Changes from baseline of glucagon AUC after 12 weeks of placebo or colesevelam treatment.
  AUC values were calculated by the trapezoid method using all results between 0 and 300 minutes
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: picograms (pg)/milliter (ml) x min
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Number analyzed (Participants) | 26 | 28
picograms (pg)/milliter (ml) x min | 4 (3) | -4 (4)
Statistical Analysis 1: Comparison: Type-2 Diabetes Mellitus Patients Treated With Colesevelam vs Type-2 Diabetes Mellitus Patients Treated With Placebo; Test type: Superiority or Other; p < 0.1, mixed-effects regression models

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Type-2 Diabetes Mellitus Patients Treated With Colesevelam | Type-2 Diabetes Mellitus Patients Treated With Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 19/26 | 23/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3.57% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type-2 Diabetes Mellitus Patients Treated With Colesevelam (N=26) | Type-2 Diabetes Mellitus Patients Treated With Placebo (N=28)
Abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Lethargic (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rapid pulse (Vascular disorders) | 1 (1) | 0 (0)
Chest pain (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes